CLINICAL TRIAL: NCT07107360
Title: Pain Neuroscience Education for Patients Undergoing Orthopaedic Surgery: Exploring Preoperative Anxiety and Improving Postoperative Recovery
Brief Title: The Effect of Pain Neuroscience Education on Preoperative Anxiety and Postoperative Recovery in Patients Scheduled for Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, SOzkan, asst. prof., Atlas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pain Neuroscience Education
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Orthopaedic Surgery; Upper Extremity
Keywords: pain neuroscience education; preoperative anxiety; recovery; orthopaedic surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Neuroscience Education Group (Experimental): received pain neuroscience education in addition to conventional preoperative education
  Interventions: Other: Pain Neuroscience Education
- Control Group (Active Comparator): received conventional preoperative education
  Interventions: Other: Conventional preoperative education

INTERVENTIONS:
Other: Pain Neuroscience Education — The study included two groups, consisting of participants who met the inclusion criteria and adhered to the procedures. Participants in the intervention group received a 20-minute Pain Neuroscience Education (PNE) session delivered face-to-face one hour prior to their scheduled surgery. The PNE focused on the biopsychosocial aspects of pain and included both theoretical and practical strategies for postoperative pain management.
  Arms: Pain Neuroscience Education Group
Other: Conventional preoperative education — Participants in the experimental group received pain neuroscience education, while participants in the control group received a booklet summarizing this education in addition to routine preoperative care.
  Arms: Control Group

SUMMARY:
This study aimed to investigate the effects of preoperative PNE on preoperative anxiety, pain-related beliefs, and postoperative functional outcomes in patients undergoing upper extremity orthopedic surgery.

DETAILED DESCRIPTION:
This study was designed as a single-blind, randomized controlled trial. It was conducted in accordance with the Declaration of Helsinki, adhering to ethical principles for medical research involving human participants. The study was completed with a total of 33 participants aged between 18 and 65 years who were scheduled for upper extremity surgery. Participants were randomly assigned to either the pain neuroscience education group or the control group.

The inclusion criteria were as follows: aged between 18 and 65 years; scheduled for upper extremity orthopedic surgery; able to communicate effectively (i.e., speaks Turkish fluently, understands verbal and written instructions, and has no speech impairments); and willing to voluntarily participate in the study.

Participants were excluded from the study if they met any of the following conditions: mental or cognitive impairments; are currently using medication for anxiety or related conditions; taking painkillers regularly; or have undergone any surgical procedures within the past year.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years
* scheduled for upper extremity orthopedic surgery; able to communicate effectively (i.e., speaks Turkish fluently,
* understands verbal and written instructions, and has no speech impairments);
* willing to voluntarily participate in the study.

Exclusion Criteria:

* any mental or cognitive impairments
* currently using medication for anxiety or related conditions
* taking painkillers regularly
* have undergone any surgical procedures within the past year.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
pain-related beliefs | Assessments were performed at two time points: one hour prior to surgery and one month after surgery.
  Pain Catastrophizing: The Pain Catastrophizing Scale (PCS) was developed in 1995 by Michael J. L. Sullivan and colleagues (Sullivan et al., 1995). The PCS is a 13-item self-report measure that assesses the extent of catastrophizing in the context of actual or anticipated pain. It conceptualizes catastrophizing as a multidimensional construct, measured across three subscales: rumination, magnification, and helplessness. Rumination refers to the tendency to focus on pain-related thoughts, helplessness reflects a perceived inability to cope with painful situations, and magnification represents an exaggerated interpretation of the threat value of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas University, Istanbul, Kagıthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol